CLINICAL TRIAL: NCT05955599
Title: Effect of Specific ACL Injury Prevention Training in Female Handball Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: University College Copenhagen (Other); University of Copenhagen (Other); Team Denmark (Other)
Responsible Party: Principal Investigator, Niels Jensby Nedergaard, Sub-Investigator, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-21030337
Record Dates: First submitted 2023-04-21; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: ACL Injury Prevention
Keywords: ACL Injuries; Age-related; Neuromuscular; Motor-Learning
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-adolescent Intervention (Experimental): 11-13 year old female handball players complete a supervised ACL injury prevention program twice a week (2 x 15 minutes) for a duration of 8 weeks. The ACL injury prevention training consists of three tracks focusing on 1) hamstring and hip external rotation strength; 2) medial hamstring activation; 3) single leg landing technique training with a special focus on knee control. The training is integrated in the players/team's normal handball practice.
  Interventions: Other: ACL Injury Prevention Training
- Pre-adolescent Control (Other): 11-13 year old female handball players complete a supervised shoulder injury prevention program twice a week (2 x 15 minutes) for a duration of 8 weeks. The shoulder injury prevention training consists of three tracks focusing on 1) external rotator cuff strength; 2) scapula stability; 3) core strength and trunk rotation. The training is integrated in the players/team's normal handball practice.
  Interventions: Other: Control - Shoulder Injury Prevention Training
- Adult Intervention (Experimental): Adult (≥18 year old) female handball players complete a supervised ACL injury prevention program twice a week (2 x 15 minutes) for a duration of 8 weeks. The ACL injury prevention training consists of three tracks focusing on 1) hamstring and hip external rotation strength; 2) medial hamstring activation; 3) single leg landing technique training with a special focus on knee control. The training is integrated in the players/team's normal handball practice.
  Interventions: Other: ACL Injury Prevention Training
- Adult Control (Other): Adult (≥18 year old) female handball players completed a supervised shoulder injury prevention program twice a week (2 x 15 minutes) for a duration of 8 weeks. The shoulder injury prevention training consists of three tracks focusing on 1) external rotator cuff strength; 2) scapula stability; 3) core strength and trunk rotation. The training is integrated in the players/team's normal handball practice.
  Interventions: Other: Control - Shoulder Injury Prevention Training

INTERVENTIONS:
Other: ACL Injury Prevention Training — Supervised ACL injury prevention training twice a week (2 x 15 minutes) over an 8-week period.
  Arms: Adult Intervention; Pre-adolescent Intervention
Other: Control - Shoulder Injury Prevention Training — Supervised shoulder injury prevention training twice a week (2 x 15 minutes) over an 8-week period.
  Arms: Adult Control; Pre-adolescent Control

SUMMARY:
The anterior Cruciate Ligament (ACL) injuries rates in female handball are high, particularly among adolescents. Therefore, the primary purpose of this randomized control trial is to explore the effects of an 8-week ACL injury prevention program on muscle activation of the medial hamstring muscles during sidecutting in female handball players.

Secondary aims are to evaluate if training effects are age-related (pre-adolescent: 11-13 year old vs. adults: ≥18 years old). The age-related comparisons Include:

1. Medial hamstring muscles activation during sidecutting;
2. Well-known biomechanical ACL injury-risk factors during high risk movements, such as cutting and landing tasks;
3. Cortical and muscular activity and functional connectivity patterns during controlled knee movements;
4. Visuomotor skill learning during a simple task involving the hamstring muscles.

ELIGIBILITY:
Inclusion Criteria:

* Female handball players playing in youth teams from the age group under 13 (11-13 years old) and adult (≥18 - 40 years old) females playing for elite u19 or senior teams in Denmark
* Have minimum 1 year of experience from playing handball
* Mental and physical skills to complete the electrophysiological and biomechanical tests

Exclusion Criteria:

* Girls/women outside the age groups listed above
* Prior surgeries to the lower limbs (e.g. ACL-reconstructions, meniscus lesions)
* Current intake of medications that include antidepressants, anxiolytics, anticonvulsants, antipsychotics, antiparkinson, hypnotics, stimulants, and/or antihistamines
* Neurological and/or psychiatric diagnoses
* Pregnant

Ages: 11 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Neuromuscular adaptations during sidecutting | Change from Baseline to Training Completion at 8 weeks. And retention 8-weeks after the prevention program was completed.
  Semitendinosus muscle pre-activity (sEMG) duirng handball specific sidecutting. Outcome measure is expressed in %MVC.during sidecutting.

SECONDARY OUTCOMES:
Changes in isometric strength | Change from Baseline to Training Completion at 8 weeks. And retention 8-weeks after the prevention program was completed.
  Peak isometric hamstring and hip external rotation strength, respectively. Outcome measure is expressed in force (Newtons).
Changes in 3D hip and knee joint angles | Change from Baseline to Training Completion at 8 weeks. And retention 8-weeks after the prevention program was completed.
  Hip and knee joint kinematic for sidecutting and single-leg landings. This include joint kinetics at initial contact and local maximum and minimums. Outcome is expressed in three-dimensional joint angles (degrees)
Changes in 3D hip and knee joint moments | Change from Baseline to Training Completion at 8 weeks. And retention 8-weeks after the prevention program was completed.
  Hip and knee joint kinetics for sidecutting and single-leg landings. Outcome is expressed in three-dimensional joint moments (M)
Changes in hamstring and quadriceps pre-activation | Change from Baseline to Training Completion at 8 weeks. And retention 8-weeks after the prevention program was completed.
  Hamstring (biceps femoris) and quadriceps (vastus lateralis and medialis) pre-activation (sEMG) during sidecutting and single-leg landings. Outcome measure is expressed in %MVC.
Visuomotor Skill Learning | Change from Baseline to Baseline +1 Day, Change from Baseline to Training Completion at 8 weeks. And retention 8-weeks after the prevention program was completed.
  Age-related differences in motor performance, skill acquisition and retention during and following visuomotor skill practice. Specific outcomes measure will be time on target (seconds per target).
Changes in shoulder sensorimoter stability | Change from Baseline to Training Completion at 8 weeks. And retention 8-weeks after the prevention program was completed.
  Shoulder sensorimoter stability measured as CoP length (mm) from force platform data.
Changes in Shoulder Rotator Cuff Strength | Change from Baseline to Training Completion at 8 weeks. And retention 8-weeks after the prevention program was completed.
  Peak isometric internal and external rotator cuff strength. Outcome measure is expressed in force (Newtons).

OTHER OUTCOMES:
Injury monitoring | Weekly for 16 weeks (from the start of the intervention to the end of the 8-week retention period)
  Type and number of injuries will be collected on a weekly basis using an electronical study-specific questionary. If injured, player's will be asked to complete a detailed questionary about the injury.
Training and match exposure | Weekly for 16 weeks (from the start of the intervention to the end of the 8-week retention period)
  Number of training and match hours will be collected on a weekly basis using an electronical study-specific questionary

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Department of Midwifery, Physiotherapy, Occupational Therapy and Psychomotor Therapy, Faculty of Health, University College Copenhagen, Copenhagen
  - Department of Nutrition, Exercise and Sports, University of Copenhagen, Copenhagen, Denmark, Copenhagen
  - Human Movement Analysis Laboratory, Department of Orthopaedic Surgery, Copenhagen University Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nedergaard NJ, Bencke J, Egholm J, Nielsen AL, Karabanov AN, Lundbye-Jensen J, Zebis MK. No Alterations in ACL Injury Risk Factors in Preadolescent Elite Female Handball Players Following an Eight-Week Targeted Training Intervention: A Randomised Controlled Trial. Transl Sports Med. 2026 Jan 2;2026:2570210. doi: 10.1155/tsm2/2570210. eCollection 2026. PMID 41522287